CLINICAL TRIAL: NCT04572230
Title: IMPACT: International Post Market Product Surveillance Study of IntrACranial Aneurysms Treated With an Endovascular Approach
Brief Title: International Post Market Surveillance Study of Intracranial Aneurysms Treated With an Endovascular Approach
Acronym: IMPACT
Status: Active, not recruiting | Type: Observational
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: CDM10001731
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-11

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Evolve EU: Selected hospitals for participation
  Interventions: Device: Endovascular treatment of intracranial aneurysms using a flow-diverting stent
- Evolve FR: All hospitals in France using the device
  Interventions: Device: Endovascular treatment of intracranial aneurysms using a flow-diverting stent

INTERVENTIONS:
Device: Endovascular treatment of intracranial aneurysms using a flow-diverting stent — The flow diverter brings about a reduction of blood flow to the aneurysm, which progresses over time into forming a stable thrombus within the aneurysm, as well as eventual aneurysm scarring and retraction. The flow diverter also acts as a scaffold for tissue growth across the neck of the aneurysm, which blocks the aneurysm from the artery blood flow.

SUMMARY:
IMPACT is an observational, post market study designed to provide an ongoing safety and performance evaluation of Stryker Neurovascular devices used for the treatment of intracranial aneurysms with an endovascular approach.

DETAILED DESCRIPTION:
IMPACT is an international, prospective, observational, multicenter, non-randomized, post market study designed to provide ongoing safety and performance evaluation on implantable devices used for the treatment of intracranial aneurysms with an endovascular approach. Data collection will also include details on adjunctive and ancillary devices used.

In addition, to gaining safety and performance data, this study will provide clinical evidence that may assist physicians in selecting an appropriate device(s) while describing treatment options used to treat patients with intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria (Evolve EU and Evolve FR):

* Subject has an intracranial aneurysm that can be treated with one of the proposed devices
* Subject age is ≥ 18 years
* Subject or subject's legally authorized representative (LAR) has signed written informed consent
* Subject is willing to comply with scheduled visits and examinations per institutional standard of care

Exclusion Criteria for (Evolve EU and Evolve FR):

* Subject is pregnant or plans to become pregnant her study participation*.
* Subject is currently enrolled in or plans to be enrolled in a concurrent drug or device study.
* Subject has a condition which will not allow him/her to comply with his/her post-procedure follow up per the institutional standard of care (medical condition, subject living abroad and unable to return for follow-up, e.g.).
* Subject has a non-target aneurysm treated within 30 days prior to study enrollment.
* Subject has a planned treatment of a non-target aneurysm in the same vascular territory during participation in the study.
* Subject target aneurysm is a ruptured intracranial aneurysm (unless ruptured at least 21 days prior the day of the index procedure)
* Subject has a target aneurysm other than saccular or fusiform intracranial aneurysms; e.g.: vertebrobasilar dolichoectasia (VBD)
* The parent vessel size does not fall within the indicated range defined by IFU
* Antiplatelet and/or anticoagulation therapy (e.g., aspirin and clopidogrel) is contraindicated for the subject
* Subject has not received dual anti-platelet agents prior to the procedure or equivalent in accordance with standard medical practice
* Subject has an active bacterial or viral infection
* The angiography demonstrates the anatomy is not appropriate for endovascular treatment, due to conditions such as:
* Severe intracranial vessel tortuosity or stenosis; and/or
* Intracranial vasospasm not responsive to medical therapy

Additional Key Exclusion Criteria (Evolve EU only):

* Subject has a non-target aneurysm treated within 30 days prior to study enrollment
* Subject has a planned treatment of a non-target aneurysm in the same vascular territory during participation in the study
* Subject has a modified Rankin Score (mRS) ≥3 at pre-procedure examination
* Subject has undergone previous stent assisted coiling or flow diverter treatment of a parent artery aneurysm near the location of the target aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have an intracranial aneurysm that the physician intends to treat with a Stryker Neurovascular device(s).
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Primary Performance Measure | 12 months
  Composite of 100% occlusion of the target aneurysm without significant parent artery stenosis per independent core lab assessment and with no target aneurysm retreatment
Primary Safety Endpoint | 12 months
  Stroke-related neurological death or Disabling stroke in the target vessel territory as adjudicated by an independent Clinical Events Committee (CEC)

SECONDARY OUTCOMES:
Secondary Performance Measures | Through 24 months
  Target aneurysm recanalization, Parent artery stenosis ≥ 50%, Target aneurysm retreatment, Target aneurysm occlusion status, Aneurysm size evaluation
Secondary Safety Endpoints | Through 24 months
  Procedural and device related serious adverse events, Any key neurological event of interest

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Kulcsár, PhD., MD, Principal Investigator — Universitätsspital Zürich, Klinik für Neuroradiologie; Jean-Christophe Gentric, PhD., MD, Principal Investigator — CHU Cavale Blanche Brest
Locations (32):
- Uniklinik Salzburg, Salzburg, Austria
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku
- France (19):
  - CHU Amiens, Amiens
  - CHRU Besançon, Besançon
  - CHU Pellegrin Bordeaux, Bordeaux
  - CHU Cavale Blanche Brest, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Henri Mondor Créteil, Créteil
  - CHU la Tronche Grenoble, La Tronche
  - CHU Lille, Lille
  - CHU Bron-Lyon, Lyon
  - CHU la Timone Marseille, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - Hospital Fondation Rothschild - Paris, Paris
  - La Pitié Salpétrière, Paris
  - NEURI, Kremlin Bicêtre, Paris
  - CHU Rennes, Rennes
  - CHU Charles Nicolle Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CHU Bretonneau Tours, Tours
- Germany (2):
  - Universitatsklinikum Augsburg A.o.R, Augsburg
  - University Hospital Knappschaftskrankenhaus Bochum, Bochum
- Italy (4):
  - AO Careggi Hospital, Florence
  - Ospedale Policlinico San Martino, Genova
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione Policlinico Universitario A. Gemelli, Rome
- Switzerland (2):
  - Inselspital Bern, Bern
  - University Hospital of Zurich, Zurich
- United Kingdom (2):
  - Queen Elizabeth Hospital, Birmingham
  - NHS Lothian, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
After completion of the 12-month primary endpoint report, and under the guidance of a physician lead publication committee, a multi-center abstract reporting the results will be prepared and may be presented at a major meeting(s). A multi-center publication may also be prepared for publication in a peer reviewed scientific journal.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After completion of the 12-month primary endpoint report
Access Criteria: A final report will be completed describing the results of all pre-specified outcomes, including negative results. The Sponsor will ensure investigators and regulatory authorities will receive the information contained in the final report.